CLINICAL TRIAL: NCT02249208
Title: Sentinel Lymph Node Biopsy With Superparamagnetic Iron Oxide vs. Standard Technique After Neoadjuvant Chemotherapy in Patients With Node-Positive Breast Cancer. A Randomized Controlled Trial.
Brief Title: Sentinel Lymph Node Biopsy With Superparamagnetic Iron Oxide for Breast Cancer Patients After Neoadjuvant Treatment.
Acronym: SENTINAC-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Sysmex España S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENTINAC-01
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sentinel Lymph Node; Neoadjuvant Chemotherapy; Clinically Node-Positive with biopsy-proven cN1; False-negative Rate
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tc+blue dye (Active Comparator): Sentinel Lymph Node (SLN) identification and resection using the standard technique of sub-areolar injection of technetium-99m (Tc-99m) and sub-areolar injection of vital blue dye before surgery.
  Interventions: Device: Tc+blue dye
- Tc+SPIO (Experimental): Sentinel Lymph Node (SLN) identification and resection using isotope technique of sub-areolar injection of technetium-99m (Tc-99m) and the magnetic technique with the sub-areolar injection of SPIO (Sienna+®), before surgery.
  Interventions: Device: Tc+SPIO
- SPIO alone (Experimental): Sentinel Lymph Node (SLN) identification and resection using the magnetic technique with the sub-areolar injection of SPIO (Sienna+®) before surgery.
  Interventions: Device: SPIO alone

INTERVENTIONS:
Device: Tc+blue dye — Sentinel Lymph Node (SLN) identification and resection using the standard technique of sub-areolar injection of technetium-99m (Tc-99m) and sub-areolar injection of vital blue dye before surgery
  Arms: Tc+blue dye
Device: Tc+SPIO — Sentinel Lymph Node (SLN) identification and resection using isotope technique of sub-areolar injection of technetium-99m (Tc-99m) and the magnetic technique with the sub-areolar injection of SPIO (Sienna+®), before surgery
  Arms: Tc+SPIO
Device: SPIO alone — Sentinel Lymph Node (SLN) identification and resection using the magnetic technique with the sub-areolar injection of SPIO (Sienna+®) before surgery
  Arms: SPIO alone

SUMMARY:
The purpose of this study is to determine the detection rate and the false negative rate of sentinel lymph node (SLN) by superparamagnetic iron oxide (SPIO) alone or in addition to radioisotope and compared to the standard method (blue and radioisotope) after neoadjuvant chemotherapy in patients with node-positive breast cancer converted to node negative after treatment by ultrasound. A randomized controlled trial.

DETAILED DESCRIPTION:
Identification of Sentinel node:

* Arm 1 (Tc+blue dye): Identification of SLN using the standard technique of sub-areolar injection of technetium-99m (Tc-99m) and vital blue dye before surgery.
* Arm 2 (Tc+SPIO): Identification of SLN using standard isotope technique of sub-areolar injection of technetium-99m (Tc-99m) before surgery and the magnetic technique with the sub-areolar injection of SPIO (Sienna+®) before surgery and detection with the SentiMag® probe. (Study)
* Arm 3 (SPIO alone): Identification of SLN using the magnetic technique with the sub-areolar injection of SPIO (Sienna+®) before surgery and detection with the SentiMag® probe. (Study)

Sentinel node's excision of radioactive and / or blue and / or magnetic (colored brown-brown), detection guided by hand probe gamma radiation, colorimetric and / or and SentiMag® paramagnetic probe.

Lymph nodes that are radioactive, blue, magnetic or palpable are considered SLNs and are resected and submitted for pathological analysis. The protocol required that at least 2 SLNs to be resected.

In all cases a completion axillary lymphadenectomy nodes dissection (ALND) will be performed after SLN biopsy. All SLNs will be excised and submitted before performing the ALND.

Characterization of the nodal status of patients with the detection rate and the false negative rate of SLN for each arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary invasive breast cancer with clinical stage T1 through T3, N1 through N2, M0 according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, seventh edition
* Completed or were planning to undergo neoadjuvant chemotherapy
* Prechemotherapy axillary nodal disease confirmed by fine-needle aspiration or core-needle biopsy
* The axilla is clinically and radiologically (by ultrasound) negative (ycN0) postchemotherapy and before surgery
* Removal of at least two SLNs
* Signed informed consent from each patient before study entry

Exclusion Criteria:

* T4 tumors, cN3 or cM1
* The axilla is clinically and radiologically (by ultrasound) positive (ycN1) postchemotherapy
* Intolerance or hypersensitivity to the compounds or iron dextran or superparamagnetic iron oxide or to vital blue dye or radioactive product.
* Chronic iron overload
* Pacemaker or other metallic implantable device in the chest wall
* Failure to submit to medical study for geographical, social or psychological
* Patient deprived of liberty or under guardianship
* Pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
False Negative Rate | 3 months
  The proportion of number of patients with a negative SLN biopsy with the number of patients with axillary lymph node metastases.

SECONDARY OUTCOMES:
Detection Rate | 3 months
  The Proportion of patients that SLNs was identified compared to total ALND patients.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel T Rubio, MD. PhD., Study Director — Hospital Universitario Vall D Hebron. Universidad Autónoma de Barcelona.
Locations (1):
- Hospital Universitario Vall D Hebron., Barcelona, Spain